CLINICAL TRIAL: NCT05418504
Title: Study of Tramadol Addiction Impact on Dental Anesthesia Success Among Algerian Males
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Doaa Mohamed Salah ElDin Diab ELBohy, Assisstant professor, Future University in Egypt
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: REC-FOPFUE-16/119
Record Dates: First submitted 2022-06-10; First posted 2022-06-14 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Dental Procedure
Keywords: Dental anesthesia; tramadol
MeSH Terms: interventions — Anesthesia, Dental

STUDY DESIGN:
Intervention Model Description: The recruited participants will then be divided into 2 groups the control group represented by dental patients who are not a tramadol addict & The study group with patients seeking dental service but also are tramadol addict.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non- Tramadol (Active Comparator): the control group represented by dental patients who are not a tramadol addict
  Interventions: Drug: Dental anesthesia
- Tramadol (Active Comparator): The study group with patients seeking dental service but also are tramadol addict.
  Interventions: Drug: Dental anesthesia

INTERVENTIONS:
Drug: Dental anesthesia — Dental anesthesia, used to do any dental procedure

SUMMARY:
Dental anesthesia is considered by far one of the main procedures in dentistry; the performance of a good dental anesthesia with a correct technique is paramount in controlling pain, facilitating the work of the dentist and gaining the confidence and cooperation of the patient

Tramadol is an FDA-approved medication for pain relief indicated mainly for moderate to severe pain, it is an opioid with 6 hours Half-Life and different dosages as 50mg, 100mg, 200mg and 300mg. Due to possible abuse and addiction potential, limitations to its use should be for pain that is refractive to other pain medication, such as non-opioid pain medication, unfortunately, the almost non-existent of censorship in Algeria and the disorderly framing made the obtain of tramadol as a medicine very easy which has led to a very alarming abuse of this drug

DETAILED DESCRIPTION:
Tramadol is an FDA-approved medication for pain relief indicated mainly for moderate to severe pain, it is an opioid with 6 hours Half-Life and different dosages as 50mg, 100mg, 200mg and 300mg. Due to possible abuse and addiction potential, limitations to its use should be for pain that is refractive to other pain medication, such as non-opioid pain medication, unfortunately, the almost non-existent of censorship in Algeria and the disorderly framing made the obtain of tramadol as a medicine very easy which has led to a very alarming abuse of this drug Meanwhile, apart from the systemic manifestations resulting from the abusive consumption of tramadol, it has become very clear that this opioid has a negative impact on the rapid and sufficient analgesic effect of dental anesthesia, it has been noticed that the anesthesia does not hold easily and the number of cartridges needed is increased, and therefore, a very particular attention must be attributed to the organization and control of its obtaining in order to limit its addiction in young people, an improvement of the care of patients must be offered according to the parameters necessary in the case of an addiction to tramadol

ELIGIBILITY:
Inclusion Criteria:

* Males
* ≥18 years
* With no comorbid conditions (HTN, Diabetes & Epilepsy)
* Tramadol addict (regular tramadol user)

Exclusion Criteria:

* Females
* ˂ 18 years
* With comorbid conditions (HTN, Diabetes & Epilepsy)
* ≥ 65 years males

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Anesthesia dose | 3 months
  Anesthesia carbols number through which both conc and dose needed in dental intervention in both arms

CONTACTS AND LOCATIONS:
Overall Officials: Doaa MS El-Bohy, PhD, Principal Investigator — FUE
Locations (2):
- Egypt (2):
  - Doaa El-Bohy, Cairo
  - Future University in egypt, Cairo